CLINICAL TRIAL: NCT04673513
Title: Cognitive Behavioral Therapy for Depression: Helping Clients Learn New Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel R. Strunk, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020B0354
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Depression
Keywords: Cognitive Behavioral Therapy; Depression; Randomized Clinical Trial; Cognitive Behavioral Skills
MeSH Terms: conditions — Depression | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Active Comparator): Cognitive behavioral therapy will be provided as described in Beck et al. (1979) and Beck (2011), with adaptations for the treatment of comorbid personality disorders as described in Beck et al. (2015).
  Interventions: Other: Psychotherapy
- Cognitive Behavioral Therapy - Skill enhanced (CBT-SE) (Active Comparator): This condition includes a variation of CBT (as provided in the other condition) with special emphasis on helping clients to develop the skills of CBT.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — In light of COVID-19 considerations, interventions are currently being provided via telehealth technology.

SUMMARY:
The purpose of this study is to compare two psychological treatments for major depressive disorder (MDD): cognitive-behavioral therapy (CBT) and CBT-Skill Enhanced (CBT-SE). CBT is well-studied, research-supported treatment for depression. CBT-SE is a variant of CBT that places greater focus on helping clients to developing the skills of CBT.

The study will enroll 150 participants with MDD. Participants will be randomized to CBT or CBT-SE, with 75 participants being assigned to each condition. For both conditions, treatment will be provided over 12 weeks, with a 6 month follow-up period.

Potential participants are asked to complete an initial screening and an intake evaluation to determine eligibility. After entering the study, participants are asked to complete evaluations at 4 weeks and at 12 weeks. They are also asked to respond to self-report instruments before and after each session. Following the 12 week treatment, participants are asked to complete monthly follow-up surveys for 6 months.

The primary objectives of this study are three-fold. The first is to compare the outcomes of the two treatments. The second is to evaluate potential mediators of any treatment differences. The third is to evaluate the process of change in these two versions of CBT.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of major depressive disorder (MDD) according to DSM-5 criteria;
2. 18 years old or older;
3. residence in the state of Ohio;
4. access to a reliable internet connection (to participate in virtual sessions); and
5. being able and willing to give informed consent.

Exclusion Criteria:

1. current or past diagnosis of bipolar disorder or a psychotic disorder;
2. moderate or severe substance use in the past 6 months (where "moderate" is defined as 4-5 symptoms and "severe" is defined as 6 + symptoms of those listed in DSM-5 for each of the substance-related disorders);
3. current disorder other than MDD if it constitutes the predominant aspect of the clinical presentation and if it requires treatment other than that being offered;
4. currently participating in a treatment for an emotional disorder, including any individual psychotherapy or psychiatric medications used to treat a mood or anxiety disorders;
5. clear indication of secondary gain (e.g., court-ordered treatment); and
6. current suicide risk or significant intentional self-harm in the last six months sufficient to preclude treatment on an outpatient basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Change in Quick Inventory of Depressive Symptoms-Self-Report at week 12. | Weeks 0-12, assessments occurred at every session through week 12.
  The Quick Inventory of Depressive Symptoms-Self-Report is a 16-item self-report measure of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depressive symptoms.
Change in Cognitive Change Sustained at week 12. | Weeks 0-12, assessments occurred at every session aside from session 1 through week 12.
  The Cognitive Change Sustained is a 9-item measure designed to assess the degree to which experienced cognitive change and used cognitive and behavioral strategies in the days leading up to their session. Scores range from 0 to 54, with a higher score indicating greater cognitive change.
Change in Ways of Responding Scale at week 12. | Weeks 0-12, assessments occurred at intake, week 4, and week 12.
  The Ways of Responding Scale is a measure of the skills taught in CBT for depression. Participants respond to 6 hypothetical stressful situations in which their initial thoughts regarding the event are given. Quality scores range from 0 to 6, with a higher score indicating greater CBT skills.
Change in CBT Skills - Interview at week 12. | Weeks 0-12, assessments occurred at intake, week 4, and week 12.
  The CBT skills interview is a semi-structured interview based measure of CBT skills. Assessors evaluate the clients CBT skills use over the past two weeks with seven items. This interview assesses client skills in using coping strategies central to CBT. Scores range from 0 to 28, with a higher score indicating greater CBT skills.

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptoms-Clinician version at week 12. | Weeks 0-12, assessments occurred at intake, week 4, and week 12.
  The Quick Inventory of Depressive Symptoms-Clinician version is a 16-item measure of depressive symptom severity. Scores range from 0 to 27, with higher scores indicating greater depressive symptoms.
Change in Cognitive Change Immediate at week 12. | Weeks 0-12, assessments occurred at every session through week 12.
  The Cognitive Change Sustained is a 5-item measure of the extent to which the client adopted new perspectives in session. It is completed following each session. Scores range from 0 to 30, with a higher score indicating greater cognitive change.
Change in Competencies of Cognitive Therapy Scale - client version at week 12. | Weeks 0-12, assessments occurred at intake, week 4, and week 12.
  The Competencies of Cognitive Therapy Scale - client version is a 29-item self-report scale that measures three areas in which clients are expected to acquire competencies from participating in CBT: behavioral activation, coping with automatic thoughts, and knowledge of schemas or core beliefs. Scores range from 29 to 203, with a higher score indicating greater CBT skills.
Change in Competencies of Cognitive Therapy Scale - therapist version at week 12. | Weeks 0-12, assessments occurred at intake, week 4, and week 12.
  The Competencies of Cognitive Therapy Scale - therapist version is a 9-item self-report scale measures three areas in which clients are expected to acquire competencies from participating in CBT: behavioral activation, coping with automatic thoughts, and knowledge of schemas or core beliefs. Scores range from 0 to 54, with a higher score indicating greater CBT skills.
Change in Work Social Adjustment Scale at week 12. | Weeks 0-12, assessments occurred at intake, week 4, and week 12.
  The Work Social Adjustment Scale is a 5-item self-report measure of functioning. Items assess the extent to which the client's functioning is impaired with regard to the client's ability to work, manage problems at home, participate in social and private leisure activities, and form close relationships. Scores range from 0 to 40, with a higher score indicating greater impairment.

OTHER OUTCOMES:
Time to relapse per modified version of the Patient Health Questionnaire | Immediately post-treatment to 6 months post treatment. Assessments occurred monthly following the posttreatment evaluation
  The Patient Health Questionnaire is a self-report measure based on the diagnostic criteria for major depressive disorder. A modified version termed the PHQ-9-H (i.e., we changed the wording in the instructions from "Over the past 2 weeks…" to "During the worst 2 weeks…") will be administered to treatment responders every month during the post-treatment follow-up period. Scores range from 0 to 27, with a higher score indicating greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Strunk, PhD, Principal Investigator — Ohio State University
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will consider requests for data sharing, pending approval from our IRB.

REFERENCES:
- [Background] Beck AT, Rush AJ, Shaw BF, Emery G. (1979). Cognitive Therapy of Depression. Guilford.

DOCUMENTS (1):
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT04673513/ICF_000.pdf